CLINICAL TRIAL: NCT01089621
Title: An Open-label Feasibility Study of Duloxetine in Adolescents With Juvenile Primary Fibromyalgia Syndrome: A Pilot Study
Brief Title: A Study for Adolescents With Fibromyalgia Syndrome
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Terminated due to study design changes; zero patients enrolled.
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12865; F1J-MC-HMGE (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-03-17; First posted 2010-03-18 (Estimated); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Duloxetine (Experimental)
  Interventions: Drug: Duloxetine

INTERVENTIONS:
Drug: Duloxetine — 30 mg to 120 mg administered orally, daily for 12 weeks
  Other Names: Cymbalta; LY248686

SUMMARY:
The purpose of this study is to evaluate the possibility of conducting a larger study in adolescents with fibromyalgia syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Meet criteria for juvenile primary fibromyalgia syndrome as defined by Yunus and Masi.
* Have a score of greater than or equal to 40mm on item 3 of the Pediatric Pain Questionnaire at screening and treatment baseline.
* Female patients must have a negative pregnancy test at baseline and must agree to abstain from sexual activity or use a reliable method of birth control.
* Patients must be capable of swallowing study drug whole.
* Patients must have venous access sufficient to allow blood sampling and be compliant with blood draws as per the protocol.

Exclusion Criteria:

* Are currently enrolled in, or discontinued within the last 30 days from, a clinical trial involving an investigational drug or device, or off-label use of a drug or device, or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study.
* Have pain symptoms related to traumatic injury, past surgery, structural bone or joint disease (such as osteoarthritis, bursitis, tendonitis), or regional pain syndrome that will interfere with the interpretation of outcome measures.
* Have a confirmed current or previous diagnosis of rheumatoid arthritis, inflammatory arthritis, or infectious arthritis, or an autoimmune disease.
* Have any primary Axis diagnosis OTHER than major depressive disorder (MDD) and/or generalized disorder (GAD) as defined by the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV), currently or within the past year. Patients with specific phobias may participate in this study.
* Have any lifetime DSM-IV Axis I diagnosis of psychosis, bipolar disorder, or schizoaffective disorder.
* Have any DSM-IV Axis II disorder which, in the judgment of the investigator, would interfere with protocol compliance.
* Have a history of substance abuse or dependence within the past year, excluding nicotine and caffeine.
* Have a positive urine drug screen for any substances of abuse or excluded medication.
* Have a family history of 1 or more first-degree relatives (parents or siblings) with diagnosed bipolar I disorder.
* Have a significant suicide attempt within 1 year of screening or are currently at suicidal risk in the opinion of the investigator.
* Have a weight less than 20 kg at any screening phase.
* Have initiated, stopped, or changed the type or intensity of psychotherapy within 3 months prior to screening.
* Have a history of seizure disorder (other than febrile seizures).
* Have abnormal thyroid-stimulating hormone (TSH) concentrations. Patients with hypothyroidism who have been treated on a stable dose of thyroid supplement for at least the past 3 months and have medically appropriate TSH concentrations, and are clinically euthyroid may participate in the study.
* Have acute liver injury or sever cirrhosis.
* Have previously taken duloxetine.
* Have a serious or unstable medical illness.
* Have initiated or discontinued hormone therapy within the previous 3 months.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2010-03 (Estimated); Primary Completion 2010-08 (Estimated); Study Completion 2010-08 (Estimated)

PRIMARY OUTCOMES:
Rate of enrollment | 6 months of enrollment
Rate of retention | 12 weeks of treatment

SECONDARY OUTCOMES:
Change in score from baseline to endpoint on the Pediatric Pain Questionnaire (PPQ) | Baseline, 12 weeks
Change in score from baseline to endpoint on the Brief Pain Inventory (BPI) modified short form severity | Baseline, 12 weeks
Change in score from baseline to endpoint on the Clinical Global Impression of Severity, overall (CGI-Severity: overall) scale | Baseline, 12 weeks
Endpoint score of Patient Global Impression of Improvement (PGI-I) scale | 12 weeks
Change in score from baseline to endpoint on the Functional Disability Inventory - child version (FDI-child) scale | Baseline, 12 weeks
Change in score from baseline to endpoint on the Functional Disability Inventory - parent version (FDI-parent) scale | Baseline, 12 weeks
Change in score from baseline to endpoint on the Clinical Global Impression of Severity for Mental Illness (CGI-mental illness) scale | Baseline, 12 weeks
Change in score from baseline to endpoint on the Children's Depression Inventory (CDI) | Baseline, 12 weeks
Change in score from baseline to endpoint on the Multidimensional Anxiety Scale for Children (MASC) | Baseline, 12 weeks
Columbia Suicide-Severity Rating Scale (CSSRS) | During 12 weeks of treatment
Change in score from baseline to endpoint on the Pediatric Quality of Life Inventory - teen report (PedsQL) | Baseline, 12 weeks
Number of patients with treatment emergent abnormal laboratory values | During 12 weeks of treatment
Change from baseline to endpoint in blood pressure | Baseline, 12 weeks
Change from baseline to endpoint in heart rate | Baseline, 12 weeks
Change from baseline to endpoint in weight | Baseline, 12 weeks
Change from baseline to endpoint in height | Baseline, 12 weeks
Number of patients with treatment emergent abnormal electrocardiogram | During 12 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (9):
- United States (9):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Phoenix, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fairfield, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Louis, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Staten Island, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Canton, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cincinnati, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oklahoma City, Oklahoma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Portland, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salt Lake City, Utah